CLINICAL TRIAL: NCT02227615
Title: Profile of Metabolites After the Intake of Mango (Mangifera Indica, l.) Var. Keitt in Humans
Brief Title: Absorption of Mango in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TexasAMU-IRB2011-0735F
Record Dates: First submitted 2014-06-04; First posted 2014-08-28 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Absorption; Chemicals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugary beverage (Placebo Comparator): Sugary beverage
  Interventions: Dietary Supplement: Sugary beverage
- Mango beverage (Experimental): Mango polyphenolics
  Interventions: Dietary Supplement: Mango polyphenolics

INTERVENTIONS:
Dietary Supplement: Mango polyphenolics — Frozen Mango (Keitt) packs provided to subjects.
  Arms: Mango beverage
Dietary Supplement: Sugary beverage — 15.7g sugar, 3.8g pectin and 0.05g citric acid was added in 100ml of the control beverage.
  Arms: Sugary beverage

SUMMARY:
The objective of this research is to characterize the urinary metabolites produced after the consumption of mango pulp in an effort to begin to characterize the bioavailability of the major group of polyphenolics in mango, ester-linked gallic acids, and to provide new insight into their in vivo physiological behavior.

DETAILED DESCRIPTION:
Eleven healthy volunteers (2 male, 9 female) who had no medical history of digestive disorders or chronic diseases participated in the 10-day mango consumption study. They were aged between 21-38 years and with a weight between 45-95 kg. Participants were asked to stop taking dietary supplements for 1 week prior to the study begin and study duration and asked to avoid excessive exercise and alcohol consumption 3 days prior to the start of the study day 1 and study day 10. Participants were also required to fill out a 72-hour nutritional report at home that detailed their food consumption over the previous 3 days leading up to the first and tenth day and were reviewed for compliance. All participants fasted from fruit and vegetables, coffee and tea one day prior to study day 1 and 10 and were asked to bring in a stool sample collected prior to consumption of mango on the first day of the study. After an overnight fast of at least 12 hours, urine collections were made (baseline) and a baseline blood draw was taken from each participant. Each participant was given 400 grams of mango to consume and urine collections were made at 0-3, 3-6, 6-8, and 8-12 hours. The volume of urine was recorded and an aliquot immediately frozen at -80°C until analysis. Blood samples were also taken at 0.5, 1, 2, 3, 4, 6, 8, and 12hrs, collected in heparinized tubes and centrifuged for 10 mins at 4000 x g, 4°C. Supernatant (plasma) was aliquoted into 2mL samples, acidified with 50 μL 85% formic acid, and immediately frozen at -80° C until analysis. Participants were given 400 grams of mango to consume daily for the next eight days and the study design was repeated again on the 10th day. After completion of the tenth day of study, stool samples were collected and immediately frozen at -20°C for microbial analysis.

ELIGIBILITY:
Inclusion Criteria:

* No medical history of digestive disorders or chronic diseases

Exclusion Criteria:

* Have medical history of digestive disorders or chronic diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the levels of metabolites of gallic acid in urine after mango intake. | 1 year
  Aliquoted urine samples were thawed and centrifuged at 13,000 x g for 10 mins at 4°C immediately prior to analysis by HPLC-MSn. All quantification of metabolites (pyrogalloyl-O-glucuronide, O-methyl-gallic acid, O-methylgallic acid-O-sulfate, O-methylpyrogalloyl-O-sulfate, pyrogalloyl-O-sulfate, deoxypyrogallol-O-sulfate, O-methylpyrogalloyl-O-sulfate) was performed in full MS and expressed as gallic acid equivalents. To standardize the concentration of metabolites for the sake of comparison across varying weights, heights, and volume of urine collected by each participant; urinary creatinine concentrations were calculated for each sample using a routine Creatinine enzyme assay kit (Sigma-Aldrich). All values are expressed as mg of standard/10 mg creatinine (mg gallic acid equivalent /10mg creatinine).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Talcott, Ph.D., Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Laboratory (ESNL) in the Department of Health and Kinesiology at Texas A&M University, College Station, Texas, United States